CLINICAL TRIAL: NCT06878547
Title: VisR Ultrasound for Noninvasively Interrogating Stromal Collagen Organization in Women as a Breast Cancer Biomarker: Evaluation of Anisotropy in Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC2449; 5R01CA281150-02 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Ultrasound screening; Ultrasound elastography; ARFI Ultrasound; VisR Ultrasound; Breast cancer diagnosis; Malignant breast lesion; Benign breast lesion; Neoadjuvant chemotherapy; Non-invasive imaging; Tissue anisotropy; Elasticity; Viscosity
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biopsy and resection samples will be retained for histopathology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Women with benign breast masses: Participants in this group will be imaged once prior to biopsy, as part of the first study arm
  Interventions: Device: Ultrasound
- Women with malignant breast masses: Participants in this group will be imaged once prior to biopsy, as part of the first study arm
  Interventions: Device: Ultrasound
- Women undergoing neoadjuvant systemic therapy (NAT): Participants in this group will be imaged once before starting NAT, once approximately midway through NAT, and once after completion of NAT, as part of the second study arm
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Non-invasive breast imaging using VisR ultrasound

SUMMARY:
Purpose: This study will evaluate how measurements of tissue stiffness, viscosity, and anisotropy using non-invasive ultrasound imaging correlate with breast tumor malignancy and response to chemotherapy.

Participants: Up to 200 women with benign or malignant breast tumors for arm 1 and up to 50 women undergoing neoadjuvant chemotherapy in the breast for arm 2 will be recruited.

Procedures (methods): The research team will use an ultrasound scanner to acquire non-invasive elastography data from the breast of each subject, testing a range of transducer rotation angles. Transducer position will be monitored using a position sensor during imaging.

DETAILED DESCRIPTION:
The purpose of the proposed research is to evaluate in vivo the feasibility of ultrasound-derived metrics for stiffness, elasticity, viscosity, and anisotropy for clinical diagnostic breast imaging. These biomarkers will be measured using novel, noninvasive ultrasound technologies under development in Dr. Gallippi's laboratory: 1) Acoustic Radiation Force Impulse (ARFI) ultrasound for interrogating tissue stiffness, 2) Viscoelastic Response (VisR) ultrasound for assessing tissue elasticity and viscosity, and 3) Dynamic Displacement Anisotropy Imaging (DDAI) for measuring tissue anisotropy. This proposed pilot study has two unblinded arms, corresponding to two aims from our NIH R01 grant.

The hypothesis of this study is that ultrasound-derived stiffness, elasticity, viscosity, and anisotropy measured in breast tissue will differ between patients with malignant and benign lesions, and between patients who are responsive versus non-responsive to neoadjuvant systemic therapy (NAT). To test these hypotheses, the research team will pursue the following specific aims from the R01 grant (specific aim #1 is being addressed by a different ongoing study, IRB #24-0122):

Aim #2: Correlate in vivo VisR outcomes to collagen fiber organization in malignant and benign breast masses and surrounding stroma in women, and demonstrate the clinical relevance of such to cancer diagnosis and staging. ARFI, VisR, and DDAI imaging will be performed on women with malignant or benign breast tumors to determine their diagnostic value in predicting malignancy. Results will be compared with histological assessment of collagen fiber organization.

Aim #3: Correlate in vivo VisR outcomes to pre- and post-NAT collagen fiber organization, and demonstrate the clinical relevance of such to predicting pathologic complete response (pCR) to NAT in women. ARFI, VisR, and DDAI imaging will be performed on women with malignant breast tumors undergoing neoadjuvant systemic therapy to monitor changes in mechanical properties during treatment and predict response to chemotherapy from early timepoints. Results will be compared with histological assessment of collagen fiber organization.

ELIGIBILITY:
Inclusion Criteria (Arm 1):

* Subjects are 20-90 years of age
* Subjects are female
* Breast lesion is sonographically visible with B-Mode ultrasound on diagnostic workup
* Breast lesion(s) have BI-RADS 4a, 4b, 4c, or 5 rating

Exclusion Criteria (Arm 1):

* Inability to provide informed consent
* Inability to communicate in English
* Inability to remain motionless for 15 minutes
* Subjects with breast implants
* Breast mass is deeper than 4 cm from skin surface
* Subjects who are pregnant or lactating
* Subjects who have pacemakers or implanted cardioverters
* Subjects with a history of mastectomy
* Previous biopsy or surgery to the site of the mass, surgical excision of mass of interest
* Subject is male

Inclusion Criteria (Arm 2):

* Subjects are 20-90 years of age
* Subjects are female
* Breast lesion is sonographically visible with B-Mode ultrasound on diagnostic workup
* Breast lesion(s) have BI-RADS 6 rating, subject will be undergoing NAT for stage 2 or 3 malignant breast lesion(s)

Exclusion Criteria (Arm 2):

* Inability to provide informed consent
* Inability to communicate in English
* Inability to remain motionless for 15 minutes
* Subjects with breast implants
* Breast mass is deeper than 4 cm from skin surface
* Subjects who are pregnant or lactating
* Subjects who have pacemakers or implanted cardioverters
* Subjects with a history of mastectomy
* Previous biopsy or surgery to the site of the mass, surgical excision of mass of interest
* Subject is male

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be patients 20-90 years of age. In the first study arm, patients with suspicious breast lesions that are rated 4 (suspicious)or 5 (highly suggestive of malignancy) on the BI-RADS scale will be recruited. In the second study arm, patients with confirmed malignant breast lesion (s) (BI-RADS 6) who are to undergo neoadjuvant systemic therapy will be recruited. All patients will be recruited from and imaged at the University of North Carolina Hospitals. Based on local demographics, we estimate that roughly 20% will be racial and ethnic minorities. Children will not be included in this study. There will be no randomization to study arms and no intervention beyond ARFI, VisR, and DDAI ultrasound imaging.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-08-25 (Estimated); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
ARFI Peak Displacement (PD) in lesion (Study Arm 1) | Baseline imaging
  Average ARFI Peak Displacement (PD) value inside of lesion. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
ARFI Peak Displacement (PD) in surrounding tissue (Study Arm 1) | Baseline imaging
  Average ARFI Peak Displacement (PD) value in an area of breast tissue outside of lesion. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
VisR Relative Elasticity (RE) in lesion (Study Arm 1) | Baseline imaging
  Average VisR RE value in lesion. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Relative Elasticity (RE) in surrounding tissue (Study Arm 1) | Baseline imaging
  Average VisR RE value in area of tissue outside of the lesion. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Relative Viscosity (RV) in lesion (Study Arm 1) | Baseline imaging
  Average VisR RV value in lesion. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Relative Viscosity (RV) in surrounding tissue (Study Arm 1) | Baseline imaging
  Average VisR RV value in area of tissue outside of the lesion. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
ARFI PD DoA in lesion (Study Arm 1) | Baseline imaging
  Ratio of maximum to minimum (DoA) of ARFI PD inside the lesion over four imaging angles
ARFI PD DoA in surrounding tissue (Study Arm 1) | Baseline imaging
  Ratio of maximum to minimum (DoA) of ARFI PD in an area of tissue outside of the lesion over four imaging angles
VisR RE DoA in lesion (Study Arm 1) | Baseline imaging
  Ratio of maximum to minimum (DoA) of VisR RE inside the lesion over four imaging angles
VisR RE DoA in surrounding tissue (Study Arm 1) | Baseline imaging
  Ratio of maximum to minimum (DoA) of VisR RE in an area of tissue outside of the lesion over four imaging angles
VisR RV DoA in lesion (Study Arm 1) | Baseline imaging
  Ratio of maximum to minimum (DoA) of VisR RV inside the lesion over four imaging angles
VisR RV DoA in surrounding tissue (Study Arm 1) | Baseline imaging
  Ratio of maximum to minimum (DoA) of VisR RV in an area of tissue outside of the lesion over four imaging angles
ARFI Peak Displacement (PD) in lesion (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Average ARFI Peak Displacement (PD) value inside of lesion. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
ARFI Peak Displacement (PD) in surrounding tissue (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Average ARFI Peak Displacement (PD) value in an area of breast tissue outside of lesion. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
VisR Relative Elasticity (RE) in lesion (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Average VisR RE value in lesion. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Relative Elasticity (RE) in surrounding tissue (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Average VisR RE value in area of tissue outside of the lesion. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Relative Viscosity (RV) in lesion (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Average VisR RV value in lesion. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Relative Viscosity (RV) in surrounding tissue (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Average VisR RV value in area of tissue outside of the lesion. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
ARFI PD DoA in lesion (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Ratio of maximum to minimum (DoA) of ARFI PD inside the lesion over four imaging angles
ARFI PD DoA in surrounding tissue (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Ratio of maximum to minimum (DoA) of ARFI PD in an area of tissue outside of the lesion over four imaging angles
VisR RE DoA in lesion (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Ratio of maximum to minimum (DoA) of VisR RE inside the lesion over four imaging angles
VisR RE DoA in surrounding tissue (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Ratio of maximum to minimum (DoA) of VisR RE in an area of tissue outside of the lesion over four imaging angles
VisR RV DoA in lesion (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Ratio of maximum to minimum (DoA) of VisR RV inside the lesion over four imaging angles
VisR RV DoA in surrounding tissue (Study Arm 2) | From enrollment to end of neoadjuvant systemic therapy, assessed up to 8 months
  Ratio of maximum to minimum (DoA) of VisR RV in an area of tissue outside of the lesion over four imaging angles

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Gallippi, PhD, Principal Investigator — Lampe Joint Department of Biomedical Engineering
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.